CLINICAL TRIAL: NCT01667302
Title: A Phase II Study of Radiotherapy Followed by Chemotherapy With DICEP Regimen in Patients With NK/T-cell Lymphoma
Brief Title: Radiotherapy Followed by Adjuvant Chemotherapy in NK/T-cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ye Guo, Assocaite Director of Medical Oncology Department, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LMTG 12-02
Record Dates: First submitted 2012-08-13; First posted 2012-08-17 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Extranodal NK/T-cell Lymphoma, Nasal Type
Keywords: NK/T-cell lymphoma; Radiotherapy; Adjuvant chemotherapy
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — Etoposide; pegaspargase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiotherapy followed by chemotherapy (Experimental): Radiotherapy Technique: IMRT Total dose: 50 Gy Per fraction: 2 Gy Chemotherapy: q3w Dexamethasone 40 mg d1-4 Ifosfamide 1200mg/m2 d1-4 Etoposide 60 mg/m2 d1-4 Cisplatin 20mg/m2 d1-4 Peg-asparaginase 2000 IU/m2 d1
  Interventions: Drug: Radiotherapy followed by chemotherapy

INTERVENTIONS:
Drug: Radiotherapy followed by chemotherapy — Radiotherapy Technique: IMRT Total dose: 50 Gy Per fraction: 2 Gy Chemotherapy: q3w Dexamethasone 40 mg d1-4 Ifosfamide 1200mg/m2 d1-4 Etoposide 60 mg/m2 d1-4 Cisplatin 20mg/m2 d1-4 Peg-asparaginase 2000 IU/m2 d1
  Other Names: DXM, IFO, VP-16, DDP, PEG-ASP

SUMMARY:
The purpose of this study is to evaluate the efficacy and tolerability of radiotherapy followed by adjuvant chemotherapy in stage I/II NK/T-cell lymphoma.

DETAILED DESCRIPTION:
For patients with stage I/II NK/T-cell lymphoma, the sequence of radiotherapy and chemotherapy is controversial. Some studies demonstrated the advantage of upfront radiotherapy. Therefore, we designed this single-arm phase II study to evaluate the efficacy and safety of radiotherapy followed by adjuvant chemotherapy with DICE regimen plus peg-asparaginase which was proved to be effective in NK/T-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Age range 14-70 years old
* Histological confirmed, previously untreated stage I/II NK/T cell lymphoma in the upper-aerodigestive tract
* ECOG performance status 0-1
* Life expectancy of more than 3 months
* Without prior history of pancreatitis
* Adequate bone marrow and organ functions

Exclusion Criteria:

* Low risk population (Definition: stage I without local invasion, B symptoms and high LDH level)
* Pregnant or lactating women
* With contraindication of steroid including uncontrolled diabetes
* Serious uncontrolled diseases and intercurrent infection
* History of other malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
3-year Progression-free survival | 3 years

SECONDARY OUTCOMES:
Overall response rate | 3 years
3-year overall survival | 3 years
Safety | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ye Guo, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Liu Y, Xue K, Xia Z, Jin J, Wang J, Sun H, Lv F, Liu X, Cao J, Hong X, Guo Y, Ma X, Zhang Q. Radiotherapy followed by DICEP regimen in treatment of newly diagnosed, stage IE/IIE, extranodal NK/T-cell lymphoma patients. Cancer Med. 2020 Aug;9(15):5400-5405. doi: 10.1002/cam4.3207. Epub 2020 Jun 9. PMID 32519518